CLINICAL TRIAL: NCT00629590
Title: A Single-Center, Open-Label, Randomized Pilot Study of the Safety and Efficacy of AzaSite® Ophthalmic Solution, 1% in Combination With Mechanical Therapy Versus Mechanical Therapy Alone for Two Weeks in Subjects With Posterior Blepharitis
Brief Title: Safety and Efficacy Pilot Study of AzaSite (Azithromycin) in Subjects With Blepharitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Inspire Pharmaceuticals, Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 041-106; P08649
Record Dates: First submitted 2008-02-21; First posted 2008-03-06 (Estimated); Last update posted 2011-09-26 (Estimated); Status verified 2011-09

CONDITIONS: Blepharitis
MeSH Terms: conditions — Blepharitis | interventions — Azithromycin

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AzaSite®
- 2 (No Intervention)

INTERVENTIONS:
Drug: AzaSite® — ophthalmic solution; 1 drop in each eye BID for two days, then 1 drop in each eye QD for ~12 days
  Other Names: AzaSite
  Arms: 1

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of AzaSite ophthalmic solution, 1% on signs and symptoms of blepharitis.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of moderate to severe chronic posterior blepharitis
* if female of childbearing potential, are non-pregnant and non-lactating

Exclusion Criteria:

* had ocular surface surgery (LASIK, refractive, etc.) within the past year
* unwilling to discontinue use of contact lenses during the study
* have glaucoma
* unable or unwilling to withhold the use of lid scrubs during the study
* have a serious systemic disease or uncontrolled medical condition that in the judgment of the investigator could confound study assessments or limit compliance
* currently using any preserved topical ocular medications (with the exception of unpreserved tear substitutes) at the time of entry into the study or during study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Change in clinical signs and symptoms associated with blepharitis | 2 weeks

SECONDARY OUTCOMES:
Standard ocular safety assessments | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Reza Haque, Study Director — works for Sponsor
Locations (1):
- South Shore Eye Care, Wantagh, New York, United States